CLINICAL TRIAL: NCT05934799
Title: An Open-label, Blinded, Randomized Crossover Four Period Single Dose Full Replicative Bioequivalence Study of Two Formulations Clopidogrel Film-coated Tablets 75 mg (Pharmtechnology LLC, Republic of Belarus) and Plavix® Film-coated Tablets 75 mg (Manufacturer: Sanofi Winthrop Industry, France; Holder RU: Sanofi-Aventis Group S.A., France) in Healthy Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Two Formulations of Clopidogrel Film-coated Tablets 75 mg in Healthy Male Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CLPDRL-CPI-2021_FRMT
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-06

CONDITIONS: Bioequivalence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other): 30 subjects assigned to the sequence TR will receive a single 75 mg dose of the test product Clopidogrel (1 x 75 mg film-coated tablet), marked as T in the sequence, in Period 1 and Period 3, and a single 75 mg dose of the reference product Plavix® (1 x 75 mg film-coated tablet), marked as R in the sequence, in period 2 and Period 4. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Clopidogrel film-coated tablet 75 mg; Drug: Plavix® film-coated tablet 75 mg
- Sequence RT (Other): 30 subjects assigned to the sequence RT will receive a single 75 mg dose of the reference product Plavix® (1 x 75 mg tablet), marked as R in the sequence, in Period 1 and Period 3 and a single 75 mg dose of the test product Clopidogrel (1 x 75 mg tablet), marked as T in the sequence, in period 2 and Period 4. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Clopidogrel film-coated tablet 75 mg; Drug: Plavix® film-coated tablet 75 mg

INTERVENTIONS:
Drug: Clopidogrel film-coated tablet 75 mg — Clopidogrel is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 75 mg of clopidogrel.
  Other Names: The test product
Drug: Plavix® film-coated tablet 75 mg — Plavix® is manufactured by Sanofi Winthrop Industry, France; holder RU: Sanofi-Aventis Group S.A., France. Each tablet contains 75 mg of clopidogrel.
  Other Names: The reference product

SUMMARY:
This is an open-labeled, randomized, four period, single-center, crossover, full replicative, comparative study, where each participant will be randomly assigned to the reference (Plavix®, 75 mg film-coated tablets) or the test (Clopidogrel, 75 mg film-coated tablets) formulation in each period of study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent.

DETAILED DESCRIPTION:
This is an open-labeled, randomized, four period, crossover, a single-center, full replicative, comparative, single-dose study, in which 60 healthy male subjects will receive one of the study treatments during each study period.

The objective of this study is to determine the bioequivalence of two different formulations of clopidogrel after a single oral dose administration under fasting conditions.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 12 hours prior to drug administration for each study period.

A subject who withdraws or is withdrawn during the pretrial evaluations but before receiving the first dose (the test or the reference product) in Period 1 will not be considered as a drop-out and will not be included in the final database. Standbys should be recruited and available to replace any subject who withdraws prior to the first drug administration. On-study drop-outs will not be replaced.

Eligible subjects will be randomized to one of two treatment sequences. There will be two sequences in the study: TR and RT, where T = the test product, R = the reference product.

For each study period, subjects will receive a single 75 mg oral dose of clopidogrel (the test or the reference formulation). Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered. For each subject, all scheduled postdose activities and assessments will be performed relative to the time of study drug administration.

Fasting will continue for at least 4 hours following drug administration, after which a standardized lunch will be served. Next meals will be provided for subjects in 6 hours, 9 hours and 12 hours after drug administration.

Water will be provided as needed until 1 hour predose. Water will be allowed beginning 2 hours after the administration of the drug.

A total of 21 blood samples will be collected (one tube of 6 mL each) in each study period for pharmacokinetic (PK) assessments. The first blood sample will be collected prior to drug administration while the others will be collected up to 24 hours after drug administration.

Сlopidogrel plasma concentrations will be measured according to a validated bioanalytical method.

Subjects are to be discharged from the clinic after the 24-hour following drug administration. However, they may be advised to stay at the clinical site for safety reasons, if judged necessary by the physician in charge.

Statistical analysis of all PK parameters will be based on an ANOVA model. Bioequivalence boundaries will be extended. The maximum extension range is 69.84%-143.19%. In order to expand the criterion of acceptability, it is necessary to confirm that the Cmax variability of the reference drug in the study actually exceeds 30%. Expansion of acceptable bioavailability limits based on intraindividual variability does not extend to AUC0-t, the limits of which, regardless of variability, should be limited to an interval of 80.00-125.00%.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy european men aged between 18 to 45 years
2. signed informed consent
3. Subjects having no clinically significant medical history and no clinically significant abnormalities in general physical examination, laboratory assessments and imaging studies
4. Body mass index 18.5-30 kg/m²
5. The results of an X-ray or fluorographic examination of the chest organs within the normal range (the results of an examination carried out within 12 months before the start of the study may be provided)
6. consent to use a double barrier method of contraception (condom + spermicide) or complete sexual abstinence, as well as consent not to participate in sperm donation during the entire study and 14 days after taking the drug in the second period.
7. Subjects are able to understand the requirements of the study, to sign a written informed consent, and also to accept all the restrictions imposed during the course of the study, and to agree to return for the required investigations.

Exclusion Criteria:

1. burdened allergic history, hypersensitivity to сlopidogrel or excipients that are part of any of the investigational drugs, or intolerance to these components;
2. clinically significant pathologies of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys and blood;
3. other diseases that, in the opinion of the researcher, may affect the absorption, distribution, metabolism or excretion of both drugs, or increase the risk of negative consequences for the volunteer;
4. the presence of mental disorders, including a history;
5. surgical interventions on the gastrointestinal tract, with the exception of appendectomy;
6. acute infectious diseases that ended less than 4 weeks before taking the drug in the first period;
7. dehydration due to diarrhea, vomiting or other reason within the last 24 hours before taking the drug in the first period of the study;
8. clinically significant abnormalities on the ECG, the level of systolic blood pressure (SBP) measured in the sitting position at the time of screening ≤ 100 mm Hg or ≥ 139 mm Hg and / or diastolic blood pressure (DBP) ≤ 70 mm Hg or ≥ 89 mm Hg;
9. heart rate less than 60 beats/min or more than 90 beats/min at the time of screening, respiratory rate less than 12 or more than 18 per minute at the time of screening, body temperature below 36.0 ° C or above 37.0 °C at the time of screening;
10. use of any drugs including herbs and food additives, vitamins that can have a significant effect on the PK of сlopidogrel or data on the effect of which on the pharmacokinetics of lisinopril are unknown, as well as question the characterization of the volunteer as healthy, less than 14 days before taking the drug in the first period;
11. increased risk of bleeding (eg, frequent nosebleeds, recent trauma, surgery, or other pathological condition);
12. a history of active pathological bleeding (eg, peptic ulcer, intracranial hemorrhage);
13. taking known inhibitors or inducers of microsomal liver enzymes, especially those affecting the CYP2C19 isoenzyme (barbiturates, omeprazole, esomeprazole, fluvoxamine, fluoxetine, moclobemide, voriconazole, fluconazole, ticlopidine, ciprofloxacin, cimetidine, carbamazepine, oxcarbazepine, chloramphenicol) or antivirals less than 2 months before taking the drug in the first period;
14. donation of plasma or blood (450 ml or more) less than 2 months (60 days) before taking the drug in the first period;
15. consumption of caffeine and xanthine-containing drinks and products (tea, coffee, chocolate, cola, etc.), products containing poppy seeds, less than 48 hours before taking the drug in the first period;
16. consumption of alcohol and alcohol-containing foods and beverages less than 48 hours before taking the drug in the first period;
17. use of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including juices, fruit drinks, etc.) less than 7 days before taking the drug in the first period;
18. intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of dry wine or 50 ml of spirits ethyl 40%) or history of alcoholism, drug addiction, drug abuse;
19. following any low-sodium diet for 2 weeks before taking drug in the first period, or following a special diet (vegetarian, vegan, with limited salt intake) or lifestyle (night work, extreme physical activity);
20. inability to refrain from intensive physical activity and contact sports less than 24 hours before taking the drug in the first period;
21. smoking more than 10 cigarettes per day less than 24 hours before taking the drug in the first period;
22. participation in other clinical trials of drugs less than 3 months before taking the drug in the first period;
23. test positive for syphilis, hepatitis B, hepatitis C or HIV at the time of screening;
24. positive test for alcohol in exhaled air at screening;
25. positive urinalysis for the content of narcotic and potent substances during screening (opiates, morphine, barbiturates, benzodiazepines, cannabinoids/marijuana);
26. the value of standard laboratory and instrumental parameters that go beyond the reference values;
27. lack of intention of volunteers to comply with the Protocol requirements throughout the course of the study and/or lack, in the opinion of the Investigator, of the volunteers' ability to understand and evaluate the information on this study as part of the informed consent form signing process, in particular regarding the expected risks and possible discomfort;
28. mental, physical and other reasons that do not allow the subject to adequately assess their behavior and correctly fulfill the conditions of the study protocol;
29. tattooing and piercing within 30 days prior to first drug administration;
30. difficulty swallowing tablets;
31. difficulty with taking blood.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Cmax of сlopidogrel in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 10 min, 15 min, 20 min, 30 min, 40 min, 50 min, 1.00, 1.15, 1.30, 2.00, 2.30, 3.00, 4.00, 6.00, 8.00, 10.00 12.00, 16.00, 24.00 hours after each drug administration.
  Maximum observed concentration in plasma.
AUC0-t of сlopidogrel in plasma after administration of the test and the reference. | Time points 0.00 (prior to each drug administration) and 10 min, 20 min, 30 min, 40 min, 50 min, 1.00, 1.15, 1.30, 2.00, 2.30, 3.00, 4.00, 6.00, 8.00, 10.00 12.00, 16.00, 24.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method.

CONTACTS AND LOCATIONS:
Locations (1):
- State Autonomous Healthcare Facility of the Yaroslavl Region "Clinical Hospital No. 2", Yaroslavl, Yaroslavl Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided